CLINICAL TRIAL: NCT00352105
Title: A Phase I/II Trial of Concurrent Chemotherapy and ZD1839 (IRESSA) With Hyperfractionated Radiation Therapy, Followed by Maintenance ZD1839 (IRESSA) for Patients With Locally Advanced Squamous Cell Head and Neck Cancer
Brief Title: Cisplatin, Fluorouracil, Iressa, and Radiation Therapy Patients With Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David Adelstein (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, David Adelstein, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCF5842; P30CA043703 (NIH); CCF-5842 (Other: Cleveland Clinic IRB); ZENECA-1839/0235
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Results first posted 2012-03-01 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Fluorouracil; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Concurrent Chemotherapy and ZD1839 (Experimental)
  Interventions: Drug: cisplatin; Drug: fluorouracil; Drug: Iressa; Radiation: hyperfractionated radiation therapy

INTERVENTIONS:
Drug: cisplatin — 20mg/m2/d IV continuous infusion x4 days
  Other Names: CDDP
Drug: fluorouracil — 1000mg.m2/d IV continuous x 4 days
  Other Names: 5FU
Drug: Iressa — 250mg/PO qd x 2 years
  Other Names: ZD1839
Radiation: hyperfractionated radiation therapy — 120cGy bid

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving cisplatin, fluorouracil, and gefitinib together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects of giving cisplatin, fluorouracil, and gefitinib together with hyperfractionated radiation therapy and to see how well they work in treating patients with locally advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Explore the activity of cisplatin, fluorouracil, gefitinib, and hyperfractionated radiotherapy, in terms of 1-year survival and 1-year distant metastatic disease control, in patients with locally advanced squamous cell carcinoma of the head and neck.

Secondary

* Explore the activity of this regimen, in terms of disease-specific survival and local control, in these patients.
* Assess the toxicity of this regimen in these patients.
* Assess the complete response rate in patients treated with this regimen.
* Assess the toxicity and tolerability of long-term maintenance with gefitinib in patients rendered disease free after this treatment regimen.

OUTLINE: Patients undergo hyperfractionated radiotherapy twice daily, 5 days a week, beginning on day 1 and continuing for 6 weeks. Patients also receive fluorouracil IV continuously over 96 hours and cisplatin IV continuously over 96 hours on days 1-4 and 22-25 and oral gefitinib beginning once daily on day 1 and continuing for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3-6 months.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary* squamous cell carcinoma of the head and neck region, excluding any of the following:

  * Nasopharynx
  * Paranasal sinuses
  * Salivary glands NOTE: *Primary site must be identified
* Locoregionally confined stage III or IV disease

  * No evidence of nodal disease below the clavicles
  * No distant hematogenous metastases (M0)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC > 3,500/mm³
* Platelet count > 100,000/mm³
* Creatinine ≤ 2.0 mg/dL
* Alkaline phosphatase < 2 times normal
* AST < 2 times normal
* Bilirubin ≤ 2.0 mg/dL
* Calcium normal
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Must not be a poor compliance risk for follow-up
* No known severe hypersensitivity to gefitinib or any excipients of this drug
* No evidence of clinically active interstitial lung disease

  * Patients with chronic, stable radiographic changes who are asymptomatic are eligible
* No unstable or uncontrolled angina, clinically apparent jaundice, or active infection
* No history of any other malignancy (except squamous cell or basal cell skin cancer or cervical carcinoma in situ) unless disease free for ≥ 5 years
* No other severe, uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)

PRIOR CONCURRENT THERAPY:

* Recovered from prior oncologic or other major surgery
* No prior definitive surgery, radiotherapy, chemotherapy, immunotherapy, or epidermal growth factor receptor inhibitors for head and neck cancer
* No investigational drugs within the past 30 days
* No concurrent CYP3A4 inducers, including any of the following:

  * Phenytoin
  * Carbamazepine
  * Rifampin
  * Phenobarbital
  * Hypericum perforatum (St. John's wort)
* Concurrent surgery allowed provided gefitinib is not administered 2 weeks before and 2 weeks after surgery
* No concurrent aminoglycoside antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-04; Primary Completion 2008-09 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Adelstein, MD, Study Chair — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients accrued between April 2003 and December 2007 from clinical facility
Groups:
- 5-FU, Cisplatin, Radiation and Iressa: Patients undergo hyperfractionated radiotherapy twice daily, 5 days a week, beginning on day 1 and continuing for 6 weeks. Patients also receive fluorouracil IN continuously over 96 hrs. and cisplatin IV continuously over 96 hrs. on days 1-3 and 22-25 and oral gefitinib beginning once daily on day 1 and continuing for up to 2 years in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | 5-FU, Cisplatin, Radiation and Iressa
Started | 60
Completed | 20
Not Completed | 40
Not completed — Death | 5
Not completed — Withdrawal by Subject | 5
Not completed — Lack of Efficacy | 9
Not completed — Adverse Event | 19
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | 5-FU, Cisplatin, Radiation and Iressa
Number analyzed (Participants) | 60
Age Continuous [Mean (Standard Deviation); unit: years] | 57 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 58
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Treated With ZD1839 With Chemotherapy and Hyperfractionated Radiation That Had a 1-year Survival
Description: To explore the activity of ZD1839 with chemotherapy and hyperfractionated radiation using 1-year survival
Time Frame: at 1 year after start of treatment
Measure: Number; unit: participants
Arm/Group | 5-FU, Cisplatin, Radiation and Iressa
Number analyzed (Participants) | 60
participants | 52 (4)

2. Secondary Outcome: Number of Participants With No Local Disease at 1 Year
Description: Number of Participants with No Local Disease at 1 Year. Local disease means that the cancer came back in the same site.
Time Frame: at 1 year after start of treatment
Population: 5 early deaths not evaluable
Measure: Number; unit: participants
Arm/Group | 5-FU, Cisplatin, Radiation and Iressa
Number analyzed (Participants) | 55
participants | 48 (3)

3. Secondary Outcome: Number of Patients With Greater Than or Equal to Mild (Grade 1) Toxicity
Description: Any toxicity greater than or equal to Grade 1= mild
Time Frame: at 1 year after start of treatment
Measure: Number; unit: participants
Arm/Group | 5-FU, Cisplatin, Radiation and Iressa
Number analyzed (Participants) | 60
participants | 60

4. Secondary Outcome: Number of Patients With a Complete Response Defined as Complete Disappearance of All Clinically Detectable Tumor.
Description: Complete response rate per RECIST Criteria (CTC V3)
Time Frame: 3 years
Population: 5 early deaths were not evaluable
Measure: Number; unit: participants
Arm/Group | 5-FU, Cisplatin, Radiation and Iressa
Number analyzed (Participants) | 55
participants | 42

5. Secondary Outcome: Number of Participants Who Completed 2 Years of Therapy
Time Frame: at 2 years after start of treatment
Measure: Number; unit: participants
Arm/Group | 5-FU, Cisplatin, Radiation and Iressa
Number analyzed (Participants) | 60
participants | 20 (7)

6. Primary Outcome: Number of Participants With No Distant Metastatic Disease at 1 Year
Description: 1-year distant metastatic disease control in patients with locally advanced squamous cell head and neck cancer. Distant disease means that cancer came back in sites outside of the head and neck.
Time Frame: 1 year
Population: 5 early deaths were not evaluable
Measure: Number; unit: participants
Arm/Group | 5-FU, Cisplatin, Radiation and Iressa
Number analyzed (Participants) | 55
participants | 54 (2)

ADVERSE EVENTS:
Time Frame: For 2 years of the study
Arm/Group | 5-FU, Cisplatin, Radiation and Iressa
Serious Adverse Events (participants affected / at risk) | 60/60
Other Adverse Events (participants affected / at risk) | 55/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5-FU, Cisplatin, Radiation and Iressa (N=60)
>= Grade 3 dysphagia (Gastrointestinal disorders) | 41
>= Grade 3 mucositis (Gastrointestinal disorders) | 52
>=Grade 3:Nausea, vomiting (Gastrointestinal disorders) | 1
Death (General disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 46
Renal Dysfunction (Renal and urinary disorders) | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5-FU, Cisplatin, Radiation and Iressa (N=60)
Grade 1-2 :Nausea, vomiting (Gastrointestinal disorders) | 52
Grade 1-2 dysphagia (Blood and lymphatic system disorders) | 18
Grade 1-2 mucositis (Gastrointestinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes